#### **Sohag University**

#### **Faculty of Medicine**

#### **Department of Ophthalmology**

# Long term evaluation of Primary Congenital Glaucoma Management in Sohag University Hospital

# **Presented by**

Dr.Ghada Fathy Mohamed Hussein M.B.B.Ch

In partial fulfillment of master degree in ophthalmology

**Under supervision of** 

**Prof.Khulood Muhammed Mahmood Sayed** 

**Professor of Ophthalmology** 

Assist.Prof.Marwa Mahmoud Abdellah

**Assistant Professor of Ophthalmology** 

Sohag University 2021

#### Introduction:

Primary congenital glaucoma is the most frequent childhood glaucoma and an Important cause of blindness(1) ,PCG due to genetically determined abnormalities in trabecular meshwork and anterior chamber angle in absence of other eye and systemic developmental problems, resulting in elevated intraocular pressure.(2)

Elevated IOP is associated with classic triad of symptoms(photophobia,epiphora and blpharospasm) wich occur due to rapid expansion of the eye causing buphthalmos(Greek"ox eye"),corneal enlargement,horizontal or oblique breaks in Descemet membrane(Haabstriae) and subsequent corneal edema and opacification.IfHaabstriae and buphthalmos are seen without elevated IOP,optic nerve cupping or corneal edema,then the patient has spontaneous arrested PCG.(2) PCG is bilateral in 65-80%.(3)

Genetic consanguinity is arisk factor. Parents of PCG patient should be aware that the chance of second child with PCG is small but real.(4)

The management of PCG is directed toward lowering and controlling the IOP and treating secondary complications such as refractive changes and amblyopia. If IOP controlled, vision in the better eye ultimately can be 20/60 or better. (5)

The treatment is surgical mainly and the medical therapy used as an adjunction to surgery, the primary goal of all surgical procedures is to eliminate the resistance to aqueous out flow caused by the anatomical anomaly in the anterior chamber angle. (6)

There are four major surgical options, angle surgeries aim to open up the drinage system of the eye either from inside (goniotomy),or the out side(trabeculotomy or viscocanalostomy). Filtrating surgeries involve making a new drinage pathway for the eye(trabeculectomy, deep sclerectomy and using glaucoma drinage devices). Cyclodestructive procedure and combined surgeries.(2)

The mainstay is angle surgery if not successful,trabeculectomy enhanced with mitomycin C or implant surgery.

Mitomycin C is an antimetabolite used during the initial stages of trabeculectomy to prevent excessive postoperative scarring and this reduce risk of failure.(7)

Ologen is a flexible bio-degradable collagen matrix of animal origin, efficacy seem to be at least similar to that of MMC with advantage of being removed in case of hypotonia and the filtration blebs are flat and vascularized without increasing risk of hypotonia, infection or bleb leak. (8)

The prognosis for children with PCG is quite variable, with some achieving good vision, while other go blind. (4) vision loss secondary to corneal scarring or optic nerve damage, and often amblyopia in asymmetrical or unilateral cases. (9)

### Aim of the work:

The purpose of the present study is evaluation of management and success rate of the cases of primary congenital glaucoma in pediatric out patient clinics at Sohag university hospital.

#### Patient and methods:

This is a retrospective, case series study of cases of primary congenital glaucoma presented to pediatric out patientclinics at Sohag university hospital for evaluation and management.

#### Inclusion criteria:

-children with operated PCG >3 month of age

#### **Exclusion criteria**

-other types of operated pediatric glaucoma

# Reviewing each patient data sheet that includes:

- -detailed history : age , sex , onset and family history.
- -examination under general anaesthesia including:
- a-Anterior segment examination:transverse corneal diameter, corneal clarity,corneal edema and presence of Haab striae.
- b-IOP measurement: the main diagnostic test, done under anaesthesia using Perkins tonometer.
- c-Gonioscopy: detect angle abnormalities to exclude secondary glaucoma.
- d-Cycloplegic refraction to look for myopia and astigmatism.
- e-Axial lenghth by A-scan ultrasonography.
- f-optic nerve evaluation by direct or indirect ophthalmoscopy attention to cup to disc ratio.
- g-B-scan if cornea dosenot allow fundus examination.
- h-Informed consent will be taken from parents of these children.
- i-Approval from the Health Research Ethics Gommittee in sohag faculty of medicine.
- j –IOP followup and vision.

## Follow-up regimen:

At different follow up period was recorded.

#### List of abbreviations:

PCG:primary congenital glaucoma.

IOP:intraocular pressure.

MMC: mitomycin C.

#### **References:**

- 1- Journal of pediatric ophthalmology and strabismus 41(5),271-288,2004.
- 2- Weinreb, R.N. Grajewski A.L., Papadopoulos M., Grigg J., Freedmans. F childhood glaucoma: the 9th consensus report of the World Glaucoms Association. Netherland: Kugler publication, 2013.
- 3- Duke-Elder S congenital Deformities. St Louis: CV mosby; 1969.548-65p.
- 4- Deluise VP, Anderson DR. Primary infantile glaucoma (congenital glaucoma). Surv Ophthalmol. 1983;28:1-18.
- 5- BiglabAW, Hiles DA-the visual results following infantile glaucoma surgery. JpediatrOphthalmol Strabismus. 1979;16(6)377-81.
- 6- J François Ophthalmological 181(2),61-73,1980.
- 7- Wilkin M,Indar A,Wormald R.Intraoperative Mitomycin C for glaucoma surgery.Cochrane Database of systematic Review 2005,Issue 4.
- 8- Cilinos, Casuccio A, Dipacef, Cagini, Ferraroll, Cillino G. Biodegradable collagen matrix implant versus Mitomycin C in trabeculectomy: five year follow up. BMC Ophthalmology (2016)16-24.
- 9- YU-Wai-mac, Arno G, Brookes J, Garcia-Feijoo J, Khaw PT, Moosajee M. primary congenital glaucoma including next generation sequencing-based approach: clinical utility gene card. Eur J Hum Genet. 2018;26(11):1713-8.